CLINICAL TRIAL: NCT00186082
Title: A Randomized Controlled Trial of the Effect of Prophylactic Antibiotics on the Infection Rate in Postpartum Third and Fourth Degree Perineal Tear Repairs
Brief Title: Antibiotics for Postpartum Third and Fourth Degree Perineal Tear Repairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Yasser Yehia El-Sayed, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 95339
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Pregnancy Complications, Infectious
MeSH Terms: conditions — Pregnancy Complications, Infectious | interventions — Cefotetan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefotetan, Cefoxitin or Clindamycin (Active Comparator)
  Interventions: Drug: Cefotetan or Cefoxitin vs placebo
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Cefotetan or Cefoxitin vs placebo

INTERVENTIONS:
Drug: Cefotetan or Cefoxitin vs placebo — Cefotetan or Cefoxitin, 1 g intravenously, or Clindamycin, 900 mg intravenously.
  Normal Saline, 100 ml intravenously for placebo arm.

SUMMARY:
This study is undertaken to find out whether prophylactic antibiotics can decrease the infection rate in third and fourth degree perineal tear repairs done in the immediate postpartum period.

DETAILED DESCRIPTION:
After obtaining consent patients who sustained third or fourth degree perineal laceration after vaginal delivery were randomly assigned to a single dose of antibiotic (cefotetan or cefoxitin, 1 g intravenously or clindamycin, 900 mg intravenously, if allergic to penicillin), or placebo (100ml normal saline) intravenously.

ELIGIBILITY:
Inclusion Criteria:

- third and fourth degree perineal laceration

Exclusion Criteria:

- chorioamnionitis, HIV positive, inflammatory bowel disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
No perineal breakdown or infection | Six weeks post partum

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Result] Duggal N, Mercado C, Daniels K, Bujor A, Caughey AB, El-Sayed YY. Antibiotic prophylaxis for prevention of postpartum perineal wound complications: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1268-73. doi: 10.1097/AOG.0b013e31816de8ad. PMID 18515507